CLINICAL TRIAL: NCT06499831
Title: 18F-FET-PET/MRI Versus Standard MRI Alone for Stereotactic RadioTherapy Planning for High Grade Brain Gliomas: A Pilot Study
Brief Title: 18F-FET-PET/MRI vs Standard MRI Alone for Stereotactic RadioTherapy Planning for High Grade Brain Gliomas
Acronym: FETSMaRT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3728
Record Dates: First submitted 2022-07-26; First posted 2024-07-15 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-06

CONDITIONS: Glioma, Malignant
Keywords: FET-PET; PET, 0-(2-18F-Fluoroethyl)-L-Tyrosine; FET; Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Intervention Model Description: This study will assess differences in management based on standard of care MRI versus intended care based on FET-PET-MRI. Changes in management will be recorded as a simulation but patients will still receive routine standard of care.
Masking Description: The radiation oncologist is blinded to result from FET-FET/MRI while planning on standard fo care MRI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Grade Glioma (Experimental): 0-(2-18F-Fluoroethyl)-L-Tyrosine (FET) PET/MRI for planning of radiation therapy of post-operative grade III/IV glioma patients
  Interventions: Diagnostic Test: 0-(2-18F-Fluoroethyl)-L-Tyrosine

INTERVENTIONS:
Diagnostic Test: 0-(2-18F-Fluoroethyl)-L-Tyrosine — 0-(2-18F-Fluoroethyl)-L-Tyrosine positron emission tomography (FET) is an amino acid agent derived from tyrosine that is able to cross the blood brain barrier. It has been studied primarily in diagnosis and detection of tumor recurrence in glioblastomas with emerging evidence for its use in brain metastases. Compared to conventional MRI, FET-PET has been shown to delineate geographically distinct tumor volume in newly diagnosed GBM suggesting the complementarity of the two modalities.
  Other Names: FET

SUMMARY:
Amino acid PET imaging for brain gliomas is gaining acceptance for the diagnosis and monitoring of disease. This is commonly performed in Europe. There is an opportunity to develop this tracer for use in Ontario, specifically for accurate delineation of disease for therapy planning and for prediction of disease recurrence, which is difficult with conventional imaging and clinical assessment techniques. The goals of this project are to develop this tracer in our local setting for use in our patients, provide evidence in the Ontario setting of its utility in addressing these unmet needs, and provide pilot evidence for future clinical trials.

Gliomas are primary malignancies of the brain. The most aggressive and common form is glioblastoma multiforme (GBM), which accounts for more than 60% of all primary brain malignancies . The standard of care for patients with glioblastoma is maximally safe resection of the enhancing tumor regions and the necrotic core followed by radiotherapy with concurrent temozolomide. MRI is widely accepted as the method of choice for treatment planning and for following these patients to predict and to detect recurrent disease.

High grade gliomas represent the most common primary brain malignancy and prognosis remains poor. The most common subtype is glioblastoma which has a 5-year survival rate of approximately 5% . Despite advances in MRI techniques, prediction and diagnosis of treatment failure remains a challenge. The result is frequent imaging mixed with uncertainty regarding the presence of viable tumor versus post-treatment effects. Furthermore, follow-up of these patients represents a high cost to the health system while symptom or disease control remains limited. A more accurate means identifying viable tumor is needed to guide management, reduce costs, and ultimately to improve patient survival and quality of life.

0-(2-18F-Fluoroethyl)-L-Tyrosine positron emission tomography (FET) is an amino acid agent derived from tyrosine that is able to cross the blood brain barrier. It has been studied primarily in diagnosis and detection of tumor recurrence in glioblastomas with emerging evidence for its use in brain metastases. Compared to conventional MRI, FET-PET has been shown to delineate geographically distinct tumor volume in newly diagnosed GBM suggesting the complementarity of the two modalities.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* High grade brain glioma (Grade 3 and 4)
* No prior radiation or systemic treatment for high grade glioma
* Planned to undergo radiation therapy with the following regimens:

  * Grade 3: 54-60 Gy over 30 fractions with temozolomide
  * Grade 3: 40Gy over 15 fractions with temozolomide
  * Grade 4: 60 Gy over 30 fractions, with or without temozolomide o Grade 4: 40 Gy over 15 fractions, with or without temozolomide
* Able to tolerate PET/MRI scan with intravenous contrast
* Willing to provide informed consent.

Exclusion Criteria:

* MRI contraindication
* Creatinine clearance < 30mL/min
* Inability to lie still for 40 minutes
* Gadolinium allergy
* Prior PET imaging
* Positive pregnancy test
* Breastfeeding
* Patient unable to follow the protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Observe recurrence/evaluate diagnostic performance of PET-FET/MRI vs MRI alone | 12 Months
  To estimate the rate of change in management due to 18F-FET-PET/MRI when used in addition to standard of care MRI.

SECONDARY OUTCOMES:
Evaluate tumor volume changes | 12 Months
  Evaluate differences in total tumor volume as defined by 18F-FET-PET versus MRI pre-operatively
Evaluate recurrence | 12 Months
  Evaluate diagnostic performance of FET-PET/MRI versus MRI alone for predicting recurrence at 12 months.
Analysis of PET Data | 12 Months
  Develop and test new MRI and PET analyses to improve recurrence prediction using machine learning and conventional statistical models

CONTACTS AND LOCATIONS:
Overall Officials: Amit Singnurkar, MD, MBA, Principal Investigator — Sunnybrook Healthcare Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT06499831/ICF_000.pdf